CLINICAL TRIAL: NCT05248061
Title: Comparison of the Effects of Platelet-Rich Plasma Supplementary Exercise and Exercise Only on Pain, Muscle Strength, Functionality, and Quality of Life in Subacromial Impingement Syndrome: A Randomized Controlled Study
Brief Title: Comparison of Platelet-Rich Plasma and Additional Exercise and Exercise Only in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Lecturer, University of Beykent
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UBeykent-3
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial Impingement Syndrome; Shoulder Rehabilitation; Platelet-Rich Plasma
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Factorial Assignment randomized controlled trial 2 groups
Who Masked: Participant
Masking Description: Patients who were diagnosed with subacromial impingement syndrome, between the ages of 45 and 65, without a history of shoulder injury other than subacromial impingement in the last 1 year and/or shoulder symptoms requiring treatment, who had not had any previous shoulder surgery and who agreed to participate in the study will be included in the study. Not meeting the inclusion criteria, a history of shoulder fracture, dislocation and/or cervical radiculopathy, presence of frozen shoulder, previous shoulder surgery, local corticosteroid injection/treatment to the shoulder joint in the last 3 months, presence of neuromuscular disease, pregnancy, history of cancer Patients with unstable angina, systemic inflammatory joint disease, conditions where exercise is contraindicated, orthopedic, rheumatic or congenital disease in the affected upper extremity, and communication problems will be excluded from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): home exercise program
  Interventions: Other: Group A
- Group B (Experimental): PRP+home exercise program
  Interventions: Other: Group A; Other: Group B

INTERVENTIONS:
Other: Group A — Wand exercises; It will be applied to increase the normal range of motion of the joint. Exercises will be performed in the directions of shoulder flexion, abduction, external and internal rotation. Objects such as a round stick, walking stick and towel can be used to assist patients during exercise.
  - *Pendulum (Codman) Exercises: These exercises will be applied in 90° flexion of the waist, with the healthy hand resting on a solid place, and turning the arm back and forth, to the sides, clockwise and counterclockwise with circular movements.
  *Capsule stretching: Auto stretching (by the patient) will be applied to the posterior region of the shoulder (capsule), pectoralis minor and upper trapezius muscles.
  *Isometric shoulder exercises Isometric exercises will be given in the directions of shoulder extension, abduction, external rotation and internal rotation.
Other: Group B — The same exercises as in Group 1 will be suitable for the participants.
  * PRP will be applied in the first session and 2 weeks later. Exercises will be started 2 days after PRP application.
  * Up to 10 cc of blood will be taken from the PRP group patients by the nurse. 25 mL of venous blood will be collected from each patient at a time, using a syringe containing 2.5 mL of the anticoagulant citrate dextrose solution. After the blood taken is transferred to the special PRP kit and centrifuged for 8 minutes at 3000 rpm, in addition to the 5-6 cc platelet-rich plasma remaining in the upper part of the kit, the entire buffy coat is injected into the syringe from the region compatible with the posterior arthroscopy portal (inferior to the acromion posterolateral bone prominence) by the physician. next, from the end point of the posterior fibers of the deltoid muscle, targeting the subacromial space) will be applied. No buffering or activating agents will be used for PRP.
  Arms: Group B

SUMMARY:
Aim: The aim of this study is to compare the effects of platelet-rich plasma application with additional exercise and only exercise application on pain, muscle strength, functionality and quality of life in subacromial impingement syndrome.

Material and Method: 56 patients who applied to the clinic with the complaint of shoulder pain and were diagnosed with Subacromial impingement syndrome between February 2022 and February 2023 will be included in the study. After giving the necessary verbal and written information about the study, the patients with informed consent will be randomized and divided into 2 groups of 28 people. The cases will be randomly divided into groups and their treatment will be done by the same researchers. Evaluation will be carried out by another investigator blinded to which group the participants belong to before and after the treatment. After the initial evaluations are completed, the 1st group will be given a home exercise program that they will apply every day for 8 weeks, and the 2nd group will be given 2 doses of PRP with an interval of 2 weeks in addition to the same exercise program. Initial evaluations of the patients will be made before the treatment and will be re-evaluated at the end of the 6th month.

Personal information with the Sociodemographic Data Form prepared by us; pain severity by Visual Analogue Scale (VAS); shoulder functionality will be evaluated with the Constant Murley Score, joint range of motion with the Universal Goniometer, muscle strength with the "Hand-held" dynamometer, and quality of life with the SF-36.

Statistical Analysis: SPSS (Statistical Package for Social Sciences) (SPSS 21.0) statistical program will be used in the statistical analysis of the data. Mann Whitney-U Test will be used to determine the difference between the efficacy of treatments. P < 0.05 will be considered statistically significant in all analyses.

DETAILED DESCRIPTION:
56 patients who applied to the clinic with the complaint of shoulder pain between February 2022 and February 2023 and were diagnosed with Subacromial impingement syndrome by the investigative orthopedist according to predetermined valid criteria will be included in the study. After giving the necessary verbal and written information about the study, the patients with informed consent will be randomized and divided into 2 groups of 28 people. The cases will be randomly divided into groups and their treatment will be done by the same researchers. The evaluation will be carried out by another investigator blinded to which group the participants belong to before and after the treatment. After the initial evaluations are completed, the 1st group will be given a home exercise program that they will apply every day for 8 weeks, and the 2nd group will be given 2 doses of PRP with an interval of 2 weeks in addition to the same exercise program. Initial evaluations of the patients will be made before the treatment and will be re-evaluated at the end of the 6th month.

Patients who were diagnosed with subacromial impingement syndrome, between the ages of 45 and 65, without a history of shoulder injury other than subacromial impingement in the last 1 year and/or shoulder symptoms requiring treatment, who had not had any previous shoulder surgery and who agreed to participate in the study will be included in the study. Not meeting the inclusion criteria, a history of shoulder fracture, dislocation and/or cervical radiculopathy, presence of frozen shoulder, previous shoulder surgery, local corticosteroid injection/treatment to the shoulder joint in the last 3 months, presence of neuromuscular disease, pregnancy, history of cancer Patients with unstable angina, systemic inflammatory joint disease, conditions where exercise is contraindicated, orthopedic, rheumatic or congenital disease in the affected upper extremity, and communication problems will be excluded from the study.

The number of our volunteers was calculated with the "G power sample size calculator". In order to be able to determine at 80% power and 0.05 significance level, when the values of the first group are taken as 7.3±0.6 and the values of the second group as 6.9±0.5 using the initial and final pain scores according to the visual analag scale at a 95% confidence interval. At least 25 volunteers should be included in each group. Despite the possibility of the participants leaving the study, 3 people will be added to each group and a total of 56 volunteers will be included in the study. Consent will be obtained from the cases with a voluntary information form.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with subacromial impingement syndrome
* Between the ages of 45-65
* No history of shoulder injury other than subacromial impingement in the last 1 year and/or no shoulder symptoms requiring treatment
* Patients who have not had any shoulder surgery before and who agreed to participate in the study

Exclusion Criteria:

* Not meeting the inclusion criteria
* History of shoulder fracture, dislocation and/or cervical radiculopathy, presence of frozen shoulder, previous shoulder surgery
* Presence of neuromuscular disease who has received local corticosteroid injection/treatment to the shoulder joint in the last 3 months
* Pregnancy, history of cancer, unstable angina, systemic inflammatory joint disease, conditions where exercise is contraindicated, presence of orthopedic, rheumatic or congenital disease in the affected upper extremity
* Patients with communication problems will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Constant Murley Score | through study completion, an average of 6 months
  Omuz fonksiyonelliğini değerlendiren, objektif ve subjektif verilere dayanan bir skorlama sistemidir. Ağrı, günlük yaşam aktiviteleri, hareket ve kuvvet parametrelerinden oluşur. Toplamda 100 puan üzerinden değerlendirilir. Puan artması hastanın kliniğinin iyi olduğunu ifade eder. Türkçe güvenilirlik ve geçerlilik çalışması yapılmıştır (Çelik D. 2016).ty.
Visual Analog Scale | through study completion, an average of 6 months
  Participants are asked to select the point where they feel their pain on a 10-centimeter (cm) horizontal line. 0 - no pain, 10 - unbearable pain. Pain conditions are evaluated separately at night, during activity and at rest.

SECONDARY OUTCOMES:
Universal Goniometry | through study completion, an average of 6 months
  Goniometric measurement is a method that is frequently used in the clinical evaluation of ROM. In addition to evaluating the range of motion of the joint, it is also used to determine functional capacity, to decide on the treatment program and to determine the effectiveness of the treatment.
"Hand-held" dynamometer | through study completion, an average of 6 months
  "Hand-held" dynamometers are accepted as a more valid method for measuring muscle strength compared to isokinetic devices due to reasons such as transportation, cost and convenience.
SF-36 | through study completion, an average of 6 months
  It was developed by Rand Corporation in 1992 to examine health-related quality of life. This scale consists of 36 questions and 8 sub-dimensions (physical and social functionality, role limitation [physical and emotional], vitality, pain and mental health). In the scale, points between 0 and 100 can be obtained from each sub-dimension. The increase in the scores obtained in the scale indicates that the health-related quality of life increases.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Study Director — University Beykent
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celik D. Turkish version of the modified Constant-Murley score and standardized test protocol: reliability and validity. Acta Orthop Traumatol Turc. 2016;50(1):69-75. doi: 10.3944/AOTT.2016.14.0354. PMID 26854052
- [Result] Reed MD, Van Nostran W. Assessing pain intensity with the visual analog scale: a plea for uniformity. J Clin Pharmacol. 2014 Mar;54(3):241-4. doi: 10.1002/jcph.250. Epub 2014 Jan 23. No abstract available. PMID 24374753
- [Result] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Result] Menek B, Tarakci D, Algun ZC. The effect of Mulligan mobilization on pain and life quality of patients with Rotator cuff syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(1):171-178. doi: 10.3233/BMR-181230. PMID 30248039
- [Result] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Balasubramaniam U, Dissanayake R, Annabell L. Efficacy of platelet-rich plasma injections in pain associated with chronic tendinopathy: A systematic review. Phys Sportsmed. 2015 Jul;43(3):253-61. doi: 10.1080/00913847.2015.1005544. Epub 2015 Jan 20. PMID 25599747
- [Result] Nejati P, Ghahremaninia A, Naderi F, Gharibzadeh S, Mazaherinezhad A. Treatment of Subacromial Impingement Syndrome: Platelet-Rich Plasma or Exercise Therapy? A Randomized Controlled Trial. Orthop J Sports Med. 2017 May 19;5(5):2325967117702366. doi: 10.1177/2325967117702366. eCollection 2017 May. PMID 28567426
- [Result] Randelli P, Arrigoni P, Ragone V, Aliprandi A, Cabitza P. Platelet rich plasma in arthroscopic rotator cuff repair: a prospective RCT study, 2-year follow-up. J Shoulder Elbow Surg. 2011 Jun;20(4):518-28. doi: 10.1016/j.jse.2011.02.008. PMID 21570659
- [Result] Roddy E, Zwierska I, Hay EM, Jowett S, Lewis M, Stevenson K, van der Windt D, Foster NE; SUPPORT trial team. Subacromial impingement syndrome and pain: protocol for a randomised controlled trial of exercise and corticosteroid injection (the SUPPORT trial). BMC Musculoskelet Disord. 2014 Mar 14;15:81. doi: 10.1186/1471-2474-15-81. PMID 24625273
- [Result] Hegedus EJ, Goode AP, Cook CE, Michener L, Myer CA, Myer DM, Wright AA. Which physical examination tests provide clinicians with the most value when examining the shoulder? Update of a systematic review with meta-analysis of individual tests. Br J Sports Med. 2012 Nov;46(14):964-78. doi: 10.1136/bjsports-2012-091066. Epub 2012 Jul 7. PMID 22773322
- [Result] Rha DW, Park GY, Kim YK, Kim MT, Lee SC. Comparison of the therapeutic effects of ultrasound-guided platelet-rich plasma injection and dry needling in rotator cuff disease: a randomized controlled trial. Clin Rehabil. 2013 Feb;27(2):113-22. doi: 10.1177/0269215512448388. Epub 2012 Oct 3. PMID 23035005
- [Result] Michener LA, Walsworth MK, Doukas WC, Murphy KP. Reliability and diagnostic accuracy of 5 physical examination tests and combination of tests for subacromial impingement. Arch Phys Med Rehabil. 2009 Nov;90(11):1898-903. doi: 10.1016/j.apmr.2009.05.015. PMID 19887215
- [Result] Say F, Gurler D, Bulbul M. Platelet-rich plasma versus steroid injection for subacromial impingement syndrome. J Orthop Surg (Hong Kong). 2016 Apr;24(1):62-6. doi: 10.1177/230949901602400115. PMID 27122515